CLINICAL TRIAL: NCT00285090
Title: Bone Mineral Density, Body Composition and Growth Following Severe Burn Injury
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of volunteers
Sponsor: Kathy Prelack, PhD, RD (Other)
Responsible Party: Sponsor-Investigator, Kathy Prelack, PhD, RD, Director of Clincal Nutrition, Shriners Hospitals for Children
Organization: Shriners Hospitals for Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-P-001850/4
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Burn; Growth; Malnutrition
Keywords: Burn Injury; Calcium; Vitamin D; Bone Mineral Density
MeSH Terms: conditions — Burns; Malnutrition | interventions — Calcium; Vitamin D; Sugars

ARMS (4):
- Early Treatment (Experimental)
  Interventions: Dietary Supplement: Calcium, Vitamin D
- LateTreatment (Experimental)
  Interventions: Dietary Supplement: Calcium,Vitamin D
- Total Treatment (Experimental)
  Interventions: Dietary Supplement: Calcium, VitaminD
- No Treatment (Placebo Comparator)
  Interventions: Other: Sugar Pill

INTERVENTIONS:
Dietary Supplement: Calcium, Vitamin D
  Arms: Early Treatment
Dietary Supplement: Calcium,Vitamin D
  Arms: LateTreatment
Dietary Supplement: Calcium, VitaminD
  Arms: Total Treatment
Other: Sugar Pill
  Arms: No Treatment

SUMMARY:
The purpose of this study is two-fold. The first is to establish that bone mineral density is diminished among children admitted to this regional burn center as compared to healthy non-burned children. The second purpose of this study is to examine the short and long-term effects of calcium and vitamin D supplementation in on bone metabolism and accrual in children who have been burned.

Specific Aims: 1) To measure bone mineral content and bone mineral density and their change during growth in convalescent burned children admitted to a regional burn center and to compare them to normal, healthy children.; 2) To measure lean body mass, fat mass, total body water in convalescent burned children admitted to a regional burn center and compare them to normal, healthy children with focus on how these components of body composition relate to indices of bone mineral content and density; 3) To identify alterations in bone metabolism and calcium and vitamin D homeostasis following burn injury and relate these to bone mineral density in burned children; 4) To test the effect of short term calcium and vitamin D supplementation on improving bone mineral density, bone mineral content, and indices of calcium and vitamin D metabolism in acutely burned children.

DETAILED DESCRIPTION:
The 60 acute patients will be randomized into 4 groups. Acute patients must be enrolled within 3 weeks of their admission to be eligible for study. Treatment is defined as provision of a supplement of 1000 mg elemental calcium with 400 IU of vitamin D daily as available in our standard hospital formulary and deemed appropriate by the pharmacist. Group 1 will take the supplement of from the day of enrollment in the study to the time of wound closure. Each group will consist of 15 patients. Upon enrollment into the study, 10 mL of blood will be obtained to measure baseline 25 and 1,25 vitamin D, parathyroid hormone, alkaline phosphatase, vitamin D binding protein, tumor necrosis factor, and IL-6 . The patients will be randomized into one of 4 groups: the early treatment group (Group 1), late treatment group (Group 2), total treatment group (Group 3) and the no treatment group (Group 4). Group 1 will take a supplement of 1000 mg calcium with 400 IU of vitamin D daily during their early acute phase of care (from the day of enrollment in the study until the time of wound closure). Group 2 will take the supplement during their rehabilitation phase of care (from the time of wound closure to the time of discharge). Group 3 will take the supplement for the entire duration of their stay (from the time of enrollment into the study to the time of discharge). Group 4 will receive no supplement. Patients who have a DXA scan of less than -2 SD units and who are in a group that is not receiving a supplement at that time (Groups 1 or 4), will begin supplementation (1000 mg calcium and 400 international units vitamin D) as part of routine care. They will remain in the study for monitoring and reporting of results. Blood levels as described above for baseline assessment will be repeated every 4 weeks for all acute patients during their initial hospital admission. At the time of wound closure, all acute patients will have their bone mineral content, bone mineral density, lean body mass, fat mass and total body water measured. This will be repeated immediately prior to discharge and at their next 2 planned reconstructive admissions (approximately 6 months to 1 year; and again at 2 years). A 10 mL blood draw to measure biochemical indices as described above will be obtained during these repeat hospital admissions as well.

ELIGIBILITY:
Inclusion Criteria for acute patients:

Patient is between ages 4 and 18 at the time of study Patients must be of Black, White or Hispanic descent Patient has sustained a 30% or greater total body surface area burn Patient is enrolled ≤ 21 days of admission to the acute unit Patient is hemodynamically stable Patient does not have a history of osteopenia Inclusion criteria for reconstructive patients Child is between ages 4 to 18 Patients have sustained a 30% or greater tbsa in the last 10 years Patients must be of Black, White or Hispanic descent Live in Northeastern USA Inclusion criteria for healthy children Child is between ages 4 to 18 Patients must be of Black, White or Hispanic descent Live in Northeastern USA Child is capable of cooperating during measurement

Exclusion Criteria for patients and healthy children:

Underlying complicating disorder that manifests in bone demineralization Patient or child is not expected to return to the hospital for additional follow-up or care

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 2 mos, 6 mos (acute), then Annual
Biochemical Indicators of Vitamin D and calcium status | every 4 weeks (acute), then annual
Growth | Annual

SECONDARY OUTCOMES:
Lean Body Mass | 2 mos, 6 mos (acute), then annual

CONTACTS AND LOCATIONS:
Overall Officials: Kathrina Prelack, PhD, Principal Investigator — Shriners Burns Hospital
Locations (1):
- Shriners Burns Hospital, Boston, Massachusetts, United States